CLINICAL TRIAL: NCT02631681
Title: Supervised Group Based Exercise for Men With Prostate Cancer on Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Peter Busch Østergren, M.D., Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProstEx
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Prostatic Neoplasms; Exercise Therapy; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Men with prostate cancer on androgen deprivation therapy (Experimental): Group based supervised combined aerobic and resistance training for 12 weeks.
  Interventions: Behavioral: Group based exercise

INTERVENTIONS:
Behavioral: Group based exercise — Supervised group based combined aerobic and resistance training for 12 weeks as part of our normal clinical practice.

SUMMARY:
Exercise intervention for men with prostate cancer on androgen deprivation therapy.

DETAILED DESCRIPTION:
The aim of the project is to investigate the effects of patient education and exercise intervention implemented in daily clinical practice for men with prostate cancer on androgen deprivation therapy

* Functional capacity
* Quality of life
* Body composition
* Blood pressure

and to assess safety of progressive resistance training for participants with bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a prostate cancer diagnosis on androgen deprivation therapy

Exclusion Criteria:

* Opioid demanding treatment for skeletal pain
* Eastern Cooperative Oncology Group performance status > 2
* Inability to perform floor and machine exercises independently

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in 30second Chair-Stand test (30s-CST) | Baseline, 12 and 24 weeks
  Test of functional capacity, measured as change
Change in Graded Cycling Test with Talk Test (GCT-TT) | Baseline, 12 and 24 weeks
  Test of functional capacity, measured as change

SECONDARY OUTCOMES:
change in QoL | Baseline, 12 and 24 weeks
  European Organisation for Research and Treatment of Cancer (EORTC) cancer and prostate specific questionnaires: EORTC QLQC-30 version 3.0 and PR25
change in Body composition | Baseline, 12 and 24 weeks
  BMI, waist and hip circumference, waist-hip ratio.
change in Bloodpressure | Baseline, 12 and 24 weeks
  Systolic and diastolic bloodpressure
Safety of exercise assessed by serious adverse events according to the FDA | Study period baseline - 24 weeks
Compliance assessed by attendance and continued exercise (yes/no) | Baseline, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Østergren, MD, Principal Investigator — Herlev and Gentofte Hospital, Faculty of Health and Medical Sciences, Copenhagen University, Denmark
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Please Select An Option Below, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ostergren P, Ragle AM, Jakobsen H, Klausen TW, Vinther A, Sonksen J. Group-based exercise in daily clinical practice to improve physical fitness in men with prostate cancer undergoing androgen deprivation therapy: study protocol. BMJ Open. 2016 Jun 29;6(6):e011460. doi: 10.1136/bmjopen-2016-011460. PMID 27357198